CLINICAL TRIAL: NCT03261739
Title: An Adaptive Design Study for the Assessment of the Safety, Tolerability, and Pharmacokinetics of RYI-018 After Repeat Dosing in Subjects With Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Safety Tolerability, and PK of RYI-018 After Repeat Dosing in Subjects With Non-Alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bird Rock Bio, Inc. (Industry)
Collaborators: ProSciento, Inc. (Industry); Perspectum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRB-018-001-US
Record Dates: First submitted 2017-08-03; First posted 2017-08-25 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: NAFLD
Keywords: NAFLD, CB1 receptor blockade, anti-CB1 monoclonal antibody
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, with 3 sequential cohorts
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RYI- 018 (Experimental): The doses of RYI-018 to be evaluated in sequential cohorts will be 0.6 mg/kg, 1.2 mg/kg, and 2.5 mg/kg.
  Interventions: Biological: RYI-018
- Placebo (Placebo Comparator): vehicle control
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RYI-018 — Anti-CB1 monoclonal antibody
  Arms: RYI- 018
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
BRB-018-001 is a multicenter, adaptive design, randomized, parallel group study to evaluate the safety, tolerability, and PK of repeat IV doses of RYI-018 in subjects with NAFLD.

DETAILED DESCRIPTION:
BRB-018-001 will be conducted as a multicenter, adaptive design, randomized, parallel group study to evaluate the safety, tolerability, and PK of repeat IV doses of RYI-018 in subjects with NAFLD. Subjects in each cohort shall be randomized to either RYI-018 or placebo as weekly injection for four weeks. The active doses of RYI-018 will be as follows: Cohort 1: 0.6 mg/kg, Cohort 2: 1.2 mg/kg, and Cohort 3: 2.5 mg/kg. Primary endpoints include safety and tolerability. Secondary endpoints include pharmacokinetics and immunogenicity.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult male or females, 18 to 65 years of age (inclusive) at the time of screening.
2. BMI ≥25.0 and ≤40.0 (kg/m2) (inclusive).
3. Liver ultrasound (or transient elastography if approved by medical monitor) which qualitatively shows fatty liver or documented history of NAFLD.
4. Liver fat percentage by MRI of approximately 10% or greater (MRI to be performed only in subjects with documented NAFLD or fatty liver by ultrasound or transient elastography if approved by medical monitor).
5. Type 2 diabetes or prediabetes.
6. Negative urine drug screen/alcohol breath test at screening.
7. Non-smokers as defined by not smoked any tobacco or nicotine-containing products within 3 months prior to screening. No current use of any nicotine containing product.

Key Exclusion Criteria:

1. Positive serologic testing for HIV, HBsAg, or HCV.
2. Have any known malignancy or history of malignancy, except for basal cell or squamous cell skin cancer that has been treated with no evidence of recurrence for at least 3 months prior to Screening.
3. Have any underlying physical or psychological medical condition that, in the opinion of the Investigator or sponsor, would make it unlikely that the subject will complete the study or is not in the subject's best interest
4. Liver function tests AST or ALT >5 x ULN at screening. One repeat test may be allowed within 7 days at the discretion of the Investigator.
5. Total bilirubin > ULN at screening except in patients with a known history of Gilbert's syndrome.
6. History or presence of alcoholism or drug abuse within the 2 years prior to the first study drug administration.
7. Administration of IP in another trial within 30 Days or 5 times the investigational drug half-life, whichever is longer, prior to the first study drug administration.
8. History of cerebrovascular event acute coronary syndrome within 6 months of screening.
9. Any history of seizures, major depression, suicidality, or unexplained syncope.
10. Subjects with other active (acute or chronic) liver disease other than NAFLD/NASH (e.g., autoimmune liver disease, viral hepatitis, genetic hemochromatosis, Wilson disease, alpha-1-antitrypsin deficiency, alcohol liver disease, drug induced liver disease).
11. Use of prescription or non-prescription weight loss medications, thiazolidinediones, investigational or approved medications for NASH, or antidepressant medications within 90 days of screening.
12. Use of insulin injections within 30 days of screening.
13. History of bariatric surgery or plans for bariatric surgery or an attempt to lose weight during study.
14. Daily alcohol intake >20 g/day for women and >30 g/day for men (on average per day), as per medical history.
15. Subjects with renal dysfunction estimated glomerular filtration rate <60 mL/min/1.73 m2.
16. HbA1c >9.5% at screening.
17. Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of adverse events | Continuous through 67 days
  Subjects will be assessed for adverse events attributable to RYI-018

SECONDARY OUTCOMES:
Time to peak serum concentration | Week 1, Week 4
  Serum concentrations after single and multiple doses of RYI-018 will be measured and the highest concentration will be identified as occurring at tmax.
Peak serum concentration | Week 1, Week 4
  Serum concentrations after single and multiple doses of RYI-018 will be measured and the highest concentration will be identified as Cmax.
Area under the serum concentration versus time curve (AUC) | Week 1, Week 4
  Serum concentrations after single and multiple doses of RYI-018 will be measured and the AUC will be calculated.
Apparent volume of distribution | Week 1, Week 4
  Serum concentrations after single and multiple doses of RYI-018 will be measured and the apparent volume of distribution, Vz, will be calculated.
Immunogenicity as determined by the concentration of serum anti-RYI-018 antibodies. | Days 8, 15, 22, 29, 36, 67
  Serum samples at multiple timepoints will be collected for quantitation of anti-RYI-018 antibodies.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - BRB Site, Chula Vista, California
  - BRB Site, Miami, Florida
  - BRB Site, Orlando, Florida
  - BRB Site, San Antonio, Texas
- BRB Site, Nedlands, Western Australia, Australia
- BRB Site, Toronto, Ontario, Canada